CLINICAL TRIAL: NCT01551355
Title: Evaluation of an Intervention to Promote Healthy Heart Habits in Pre-School Children
Brief Title: Promoting Heart Health in Preschool Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valentin Fuster (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Fundación Cardioinfantil Instituto de Cardiología (Other); Sesame Workshop (Unknown)
Responsible Party: Sponsor-Investigator, Valentin Fuster, Physician-in-Chief, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: GCO 09-0702
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Health
Keywords: behavioral modification; health communication; prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children-Multicomponent intervention (Experimental): The intervened children were provided classroom educational and playful activities during 5 months, which included Sesame Workshop Healthy Habits storybooks, posters, videos, games, and songs (1 hour daily); a "Healthy family day" workshop (1 hour); and weekly health notes. Parents participated in 3 workshops and weekly notes containing positive health messages about nutrition and active lifestyles to share with their children. Teachers also participated in 3 centralized training sessions, plus personalized working sessions with a research supervisor (2 hours every 15 days), and received a teacher's guide.
  Interventions: Behavioral: Children-Multicomponent intervention
- children - control group (No Intervention): The control preschool facilities continued with their usual preschool curriculum

INTERVENTIONS:
Behavioral: Children-Multicomponent intervention — The intervened children were provided classroom educational and playful activities during 5 months, which included Sesame Workshop Healthy Habits storybooks, posters, videos, games, and songs (1 hour daily); a "Healthy family day" workshop (1 hour); and weekly health notes. Parents participated in 3 workshops and weekly notes containing positive health messages about nutrition and active lifestyles to share with their children. Teachers also participated in 3 centralized training sessions, plus personalized working sessions with a research supervisor (2 hours every 15 days), and received a teacher's guide.
  Arms: Children-Multicomponent intervention

SUMMARY:
As part of the Colombian Hearty Health Initiative program led by Mount Sinai Cardiovascular Institute, a multidisciplinary team design and implemented a pedagogic and communication strategies for the promotion of healthy heart habits (PPHH) in preschoolers. This included educational materials, pedagogical activities and the use of Sesame Workshop healthy habits for life materials. For Colombia, the latter were largely developed in collaboration with the Colombian Society of Pediatrics, Colombian Society of Cardiology and Cardiovascular Surgery, Colsubsidio and Fundación Cardioinfantil-Instituto de Cardiología.

DETAILED DESCRIPTION:
Background Increased levels of risk factors during childhood create an important life-long burden that favors the development of cardiovascular (CVD) disease in adulthood. Epidemiologic studies have demonstrated that cardiovascular disease risk factors are identifiable in childhood and persist through to adulthood. It is unknown whether interventions targeting preschoolers may change knowledge, attitudes and habits (KAH) towards healthy lifestyles and, eventually, reduce the burden of CVD.

The goal of the proposed study is to assess over a five month intervention period, the impact of an educational intervention on preschooler's knowledge of, habits and attitudes towards healthy eating and living an active lifestyle. The impact of the intervention will be also assessed in parents and teachers.

Methods The investigators will conduct a cluster, randomized controlled trial in 1216 pre-school children 3 to 5 years of age, 928 parents, and 120 teachers from 14 preschool facilities in Bogotá, Colombia in a low socioeconomic and underprivileged community. Randomization will occur at the facility level. The intervention will include classroom activities and use of printed material (books, posters, teachers' guides, games) and videos. Meanwhile, children in the control facilities will continue with their usual curriculum. A structured survey will be used at baseline and end of study to evaluate changes in KAH and the authors a priori give differential weights (70-20-10, respectively) to the scores to compose a standardized weighted total score (WTS). The primary outcome will be the change in children's WTS and the secondary outcomes will be the changes in parents' and teachers´ WTS.

Potential Impact of the Trial If found to be effective in improving the short-term changes in knowledge, attitudes and habits, the educational intervention may have the potential to influence the children's' diet and physical activity patterns throughout their lifetimes by early interventions when attitudes and habits are formed. The program also targets parents and teachers who contribute to shape children's attitudes and habits and who are often at high risk for health problems associated with unhealthy diet and limited physical activity themselves. The program aims to empower local partners in the health, education, media and government sectors to build up the capacities to ensure sustainability. If proven efficacious in the short term, further evaluative studies should test the hypothesis that this program will serve as an effective and sustainable model to improve children's health worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Children attending one of the 14 H.I. in Usaquén
* Children who are 3, 4, or 5 years of age at the time of the beginning of the intervention

Exclusion Criteria:

* Unwillingness to provide informed consent
* Children who have received formal training in healthy habits in nutrition and / or physical activity in the 6 months prior to the start of the follow-up period of the study.
* Children who plan to receive formal training in healthy habits in nutrition and / or physical activity during the follow-up study period.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2279 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, PhD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Fundación CardioInfantil Instituto de Cardiología, Bogotá, Colombia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in 14 preschool facilities in Usaquén (Bogotá, Colombia) between May and November, 2009
Groups:
- Healthy Habits Intervention: Preschool Facility* Intervention Arm children provided classroom educational and playful activities during 5 months, which included Sesame Workshop Healthy Habits storybooks, posters, videos, games, and songs (1 hour daily); a "Healthy family day" workshop (1 hour); and weekly health notes.
- Usual Curriculum: children - education imparted by teachers control preschool facilities continued with their usual preschool curriculum
- Healthy Habits Intervention - Parents/Caregivers: Parents participated in 3 workshops and weekly notes containing positive health messages about nutrition and active lifestyles to share with their children.
- Usual Curriculum - Parents/Caregivers; Usual Curriculum - Teachers: Control preschool facilities continued with their usual preschool curriculum
- Healthy Habits Intervention - Teachers: Teachers participated in 3 centralized training sessions, plus personalized working sessions with a research supervisor (2 hours every 15 days), and received teacher's guide.
Period: Overall Study
Arm/Group | Healthy Habits Intervention | Usual Curriculum | Healthy Habits Intervention - Parents/Caregivers | Usual Curriculum - Parents/Caregivers | Healthy Habits Intervention - Teachers | Usual Curriculum - Teachers
Started | 622 | 594 | 493 | 435 | 64 | 71
Completed | 571 | 545 | 459 | 411 | 55 | 65
Not Completed | 51 | 49 | 34 | 24 | 9 | 6
Not completed — Lost to Follow-up | 51 | 49 | 34 | 24 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Healthy Habits Intervention - Children: Preschool Facility* Intervention Arm children provided classroom educational and playful activities during 5 months, which included Sesame Workshop Healthy Habits storybooks, posters, videos, games, and songs (1 hour daily); a "Healthy family day" workshop (1 hour); and weekly health notes.
- Usual Curriculum - Children; Usual Curriculum - Parents/Caregivers; Usual Curriculum - Teachers: Control preschool facilities continued with their usual preschool curriculum
- Total: Total of all reporting groups
Arm/Group | Healthy Habits Intervention - Children | Usual Curriculum - Children | Healthy Habits Intervention - Parents/Caregivers | Usual Curriculum - Parents/Caregivers | Healthy Habits Intervention - Teachers | Usual Curriculum - Teachers | Total
Number analyzed (Participants) | 622 | 594 | 493 | 435 | 64 | 71 | 2279
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — not analyzed | NA (NA) — not analyzed | 31.25 (8.1) | 29.94 (6.8) | 39.04 (10.6) | 35.05 (8.9) | NA (NA) — not analyzed
Age, Customized [Number; unit: participants]
  age 3 | 342 | 309 | NA — adults | NA — adults | NA — adults | NA — adults | 651
  age 4 | 270 | 266 | NA — adults | NA — adults | NA — adults | NA — adults | 536
  age 5 | 10 | 19 | NA — adults | NA — adults | NA — adults | NA — adults | 29
Gender [Count of Participants; unit: Participants] — Children: gender (male/female)
  Participants
    Female | 296 | 275 | 412 | 373 | 55 | 64 | 1475
    Male | 326 | 319 | 81 | 62 | 9 | 7 | 804
Region of Enrollment [Number; unit: participants]
  Colombia | 622 | 594 | 493 | 435 | 64 | 71 | 2279

OUTCOME MEASURES:

1. Primary Outcome: Change in KAH Score for Children
Description: Change in weighted knowledge, attitude, habit (KAH) (70/20/10) score among children after 5 months of intervention as compared to prior to intervention.
  The study hypothesized that the mean change in knowledge scores associated with this short intervention period would be larger than the mean changes in scores due to attitudes and habits, differential weights (70, 20, and 10, respectively) were given to the scores a priori to compose a standardized weighted total score (WTS).
  The developed questionnaires measured knowledge, attitudes, and habits on healthy eating and living an active lifestyle in children, parents, and teachers.
  Scale range: 0-100 Knowledge scale range: 0-100 Attitude scale range: 0-100 Habit scale range: 0-100 WTS (weighted total score) scale range: 0-100
  Higher values represent a better outcome
Time Frame: at baseline and at 6 months
Population: The analysis was done with children that answered al questions in 3 topics: knowledge, attitudes and habits.
  Change Score in Weighted total score controlling for Cluster Effect, Sex, Age, Children's Weight, and Teacher's Educational Level after 5-Month Intervention.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Healthy Habits Intervention: Preschool Facility* Intervention Arm classroom educational and playful activities during 5 months, which included Sesame Workshop Healthy Habits storybooks, posters, videos, games, and songs (1 hour daily); a "Healthy family day" workshop (1 hour); and weekly health notes.
- Usual Curriculum: education imparted by teachers control preschool facilities continued with their usual preschool curriculum
Arm/Group | Healthy Habits Intervention | Usual Curriculum
Number analyzed (Participants) | 433 | 425
units on a scale | 7.66 [6.94 to 8.38] | 3.76 [3.4 to 4.12]
Statistical Analysis 1: Comparison: Healthy Habits Intervention vs Usual Curriculum; Test type: Superiority or Other; p < .001, t-test, 2 sided; The intervention was evaluated using generalized estimating equation models, controlling for cluster effect, sex, age, weight, and education level; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [1.64 to 6.16]

2. Secondary Outcome: KAH Score for Parents
Description: Change in Weighted knowledge, attitude, habit (KAH) score (70/20/10) among parents after 5 months of intervention as compared to prior to intervention.
  Because we hypothesized that the mean change in knowledge scores associated with this short intervention period would be larger than the mean changes in scores due to attitudes and habits, we a priori gave differential weights (70, 20, and 10, respectively) to the scores to compose a standardized weighted total score (WTS).
  Questionnaires were developedheae to measure knowledge, attitudes, and habits on healthy eating and living an active lifestyle in children, parents, and teachers.
  Scale range: 0-100 Knowledge scale range: 0-100 Attitude scale range: 0-100 Habit scale range: 0-100 WTS (weighted total score) scale range: 0-100 Higher values represent a better outcome
Time Frame: at baseline and at 6 months
Population: Change in weighted total score controlling for Cluster Effect, Sex, Age, Children's Weight, and Teacher's Educational Level after 5-Month Intervention. Data available only for 402 parents in healthy habits arm and 360 parents in usual curriculum arm.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Healthy Habits Intervention | Usual Curriculum
Number analyzed (Participants) | 402 | 360
units on a scale | 6.12 [5.53 to 6.71] | 2.04 [1.83 to 2.25]
Statistical Analysis 1: Comparison: Healthy Habits Intervention vs Usual Curriculum; Test type: Superiority or Other; p < .001, t-test, 2 sided; Mean Difference (Final Values) = 4.08, 95% CI 2-sided [2.03 to 6.12]

3. Secondary Outcome: KAH Score for Teachers
Description: Change in Weighted knowledge, attitude, habit (KAH) score (70/20/10) among teachers after 5 months of intervention as compared to prior to intervention.
  Because we hypothesized that the mean change in knowledge scores associated with this short intervention period would be larger than the mean changes in scores due to attitudes and habits, we a priori gave differential weights (70, 20, and 10, respectively) to the scores to compose a standardized weighted total score (WTS).
  We developed questionnaires to measure knowledge, attitudes, and habits on healthy eating and living an active lifestyle in children, parents, and teachers.
  Scale range: 0-100 Knowledge scale range: 0-100 Attitude scale range: 0-100 Habit scale range: 0-100 WTS (weighted total score) scale range: 0-100 Higher values represent a better outcome
Time Frame: at baseline and at 6 months
Population: Change in weighted total score controlling for Cluster Effect, Sex, Age, Children's Weight, and Teacher's Educational Level after 5-Month Intervention. Data available only for 37 teachers in healthy habits arm and 35 teachers in usual curriculum arm.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Healthy Habits Intervention | Usual Curriculum
Number analyzed (Participants) | 37 | 35
units on a scale | 7.24 [4.83 to 9.65] | 1.88 [1.23 to 2.53]
Statistical Analysis 1: Comparison: Healthy Habits Intervention vs Usual Curriculum; Test type: Superiority or Other; p = .06, t-test, 2 sided; Mean Difference (Final Values) = 5.36, 95% CI 2-sided [-0.29 to 11.01]

4. Secondary Outcome: Body Mass Index - BMI
Description: The body mass index (BMI), or Quetelet index, is a measure of relative weight based on an individual's mass and height = Kg/m²
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Kg/m²
Arm/Group | Healthy Habits Intervention | Usual Curriculum
Number analyzed (Participants) | 622 | 594
Kg/m² | 16.57 (0.45) | 16.4 (0.49)

ADVERSE EVENTS:
Description: adverse events information not collected
Arm/Group | Healthy Habits Intervention | Usual Curriculum
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
minimal participation of teachers in initial planning stage. small number of teachers evaluated has limited the statistical power in this group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes